CLINICAL TRIAL: NCT07279597
Title: An Open, Single-arm Clinical Study on the Efficacy and Safety of Toripalimab Combined With RC48-ADC in Radiotherapy for HER-2 Positive Muscle-invasive Bladder Cancer (MIBC) Patients for Bladder Preservation Treatment After Chemotherapy Induction
Brief Title: A Phase II Study of Toripalimab Plus RC48-ADC With Radiotherapy for Bladder Preservation in HER2-Positive Muscle-Invasive Bladder Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, bo liu, associate chief physician, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TongjiHospital
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Muscle-invasive Bladder Urothelial Carcinoma
Keywords: Bladder-preserving
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): This is a prospective, open-label, single-center, single-arm clinical study. Plans to enroll 45 MIBC patients with clinical stage T2-T4aN0M0 and HER2-positive (IHC 1+/2+/3+) status. Treatment Flow: Post maximal Transurethral Resection of Bladder Tumor (TURBT); 2 cycles of Gemcitabine + Cisplatin chemotherapy; 4 cycles of RC48-ADC + Toripalimab targeted therapy; Radiotherapy (60-64 Gy) with concurrent Toripalimab treatment; Continue with 6 cycles of RC48-ADC + Toripalimab after radiotherapy completion; Patients achieving CR will receive maintenance therapy with Toripalimab for 1 year.
  Interventions: Drug: RC48-ADC + Toripalimab

INTERVENTIONS:
Drug: RC48-ADC + Toripalimab — Treatment Flow: Post maximal Transurethral Resection of Bladder Tumor (TURBT); 2 cycles of Gemcitabine + Cisplatin chemotherapy; 4 cycles of RC48-ADC + Toripalimab targeted therapy; Radiotherapy (60-64 Gy) with concurrent Toripalimab treatment; Continue with 6 cycles of RC48-ADC + Toripalimab after radiotherapy completion; Patients achieving CR will receive maintenance therapy with Toripalimab for 1 year.

SUMMARY:
This is a prospective, open-label, single-center, single-arm clinical study. Plans to enroll 45 MIBC patients with clinical stage T2-T4aN0M0 and HER2-positive (IHC 1+/2+/3+) status. Treatment Flow: Post maximal Transurethral Resection of Bladder Tumor (TURBT); 2 cycles of Gemcitabine + Cisplatin chemotherapy; 4 cycles of RC48-ADC + Toripalimab targeted therapy; Radiotherapy (60-64 Gy) with concurrent Toripalimab treatment; Continue with 6 cycles of RC48-ADC + Toripalimab after radiotherapy completion; Patients achieving CR will receive maintenance therapy with Toripalimab for 1 year.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-center, single-arm clinical study. Plans to enroll 45 MIBC patients with clinical stage T2-T4aN0M0 and HER2-positive (IHC 1+/2+/3+) status. Treatment Flow: Post maximal Transurethral Resection of Bladder Tumor (TURBT); 2 cycles of Gemcitabine + Cisplatin chemotherapy; 4 cycles of RC48-ADC + Toripalimab targeted therapy; Radiotherapy (60-64 Gy) with concurrent Toripalimab treatment; Continue with 6 cycles of RC48-ADC + Toripalimab after radiotherapy completion; Patients achieving CR will receive maintenance therapy with Toripalimab for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria are eligible to participate in the trial:

  1. Male or female ≥18 years of age;
  2. ECOG Performance Status: 0-1;
  3. Patients must have undergone pathological biopsy and imaging diagnosis, and be judged by the investigator to have muscle-invasive bladder urothelial carcinoma (urothelial carcinoma as the main pathological component >50%);
  4. Clinical stage T2-T4a N0 M0 (CT/MRI ± PET/CT);
  5. HER2 immunohistochemistry 1+, 2+, or 3+;
  6. Expected survival ≥3 months;
  7. Normal function of major organs (within 14 days before enrollment), meeting the following standards:

  <!-- -->

  1. Hematological criteria must be met (no blood transfusion or granulocyte colony-stimulating factor treatment within 14 days before enrollment):

     HB ≥90 g/L; ANC ≥1.5×10^9 /L; PLT ≥100×10^9 /L;
  2. No functional organic disease, meeting the following standards:

T-BIL ≤1.5×ULN (Upper Limit of Normal); ALT and AST ≤2.5×ULN; if liver metastases are present, then ALT and AST ≤5×ULN; Serum creatinine ≤ 2×ULN, or creatinine clearance >30 ml/min (Cockcroft-Gault formula);International Normalized Ratio (INR), Activated Partial Thromboplastin Time (aPTT): ≤1.5× ULN (this criterion applies only to patients not receiving anticoagulant therapy; patients receiving anticoagulant therapy should have their anticoagulant within the therapeutic range); 8. No systemic corticosteroid treatment within 4 weeks prior to therapy; 9. Men of reproductive potential or women with childbearing potential must use highly effective contraception methods (e.g., oral contraceptives, intrauterine device, sexual abstinence, or barrier contraception combined with spermicide) during the trial and continue contraception for 12 months after the end of treatment; 10. Women with childbearing potential must have a negative urine pregnancy test result within 7 days before treatment; 11. Subjects voluntarily join the study, sign the informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Patients presenting with any of the following conditions will be excluded from the trial:

  1. Previous treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 therapy, including during the adjuvant therapy phase;
  2. Known allergy to recombinant humanized anti-PD-1 monoclonal antibody drugs or their components;
  3. Received other anti-tumor therapy (including corticosteroid therapy, immunotherapy) or participated in other clinical studies within 4 weeks before the start of study treatment, or have not recovered from previous toxicity (except for Grade 2 alopecia and Grade 1 neurotoxicity);
  4. Pregnant or lactating women;
  5. Positive HIV test result;
  6. Patients with active Hepatitis B or Hepatitis C: HBsAg or HBcAb positive with concurrently positive HBV DNA copy number (quantitative detection limit of 500 IU/ml, or reaching the positive copy number value detected by the research center); HBV DNA must be tested during study screening for these patients; Patients with positive HCV antibody test results can only be enrolled in this study if the PCR test result for HCV RNA is negative.
  7. History of definite active tuberculosis;
  8. Active autoimmune disease requiring systemic treatment in the past 2 years (e.g., using disease-modifying drugs, corticosteroids, or immunosuppressive drugs). Related replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement for renal or pituitary insufficiency) is allowed;
  9. Other severe, uncontrolled concomitant diseases that may affect protocol compliance or interfere with result interpretation, including active opportunistic infections or advanced (severe) infections, uncontrolled diabetes, cardiovascular diseases (Class III or IV heart failure as defined by the New York Heart Association classification, second-degree or higher heart block, myocardial infarction within the past 6 months, unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc.) or pulmonary diseases (interstitial pneumonia, obstructive pulmonary disease, and history of symptomatic bronchospasm);
  10. Received live vaccination within 4 weeks before the start of treatment;
  11. Previous allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
  12. Underwent major surgical procedures (excluding diagnostic surgery) within 4 weeks before the start of treatment;
  13. History of psychotropic drug abuse and inability to abstain, or history of mental disorders;
  14. Presence of clinically symptomatic large pleural effusion or ascites requiring symptomatic treatment;
  15. History of other malignancies within the past 5 years that have not been cured, excluding malignancies that are considered clearly cured or curable cancers, such as basal cell or squamous cell skin cancer, localized low-risk prostate cancer, carcinoma in situ of the cervix, or carcinoma in situ of the breast; Note: Localized low-risk prostate cancer (defined as stage ≤T2b, Gleason score ≤7, and PSA ≤20 ng/mL at diagnosis if measured) treated with curative intent and without biochemical recurrence of prostate-specific antigen (PSA) may participate in this study;
  16. Concurrent upper urinary tract urothelial carcinoma (renal pelvis, ureter urothelial carcinoma);
  17. Other severe, acute, or chronic medical or psychiatric conditions or laboratory abnormalities that, in the investigator's opinion, may increase the risk associated with study participation or may interfere with the interpretation of study results.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | Complete Response (CR) rate at 3 months after radiotherapy completion
  Complete Response (CR) rate at 3 months after radiotherapy completion (defined as: no visible tumor on imaging, negative pathological assessment from diagnostic TURBT at the tumor site, and negative urine FISH test in the Intent-to-Treat (ITT) population).

IPD SHARING:
Plan to Share IPD: No